CLINICAL TRIAL: NCT07063680
Title: Efficacy of Early Argipressin (Arginine Vasopressin) in the Management of Intensive Care Patients With Norepinephrine-refractory Vasoplegic Shock: a Multicentric Randomized, Double-blind Placebo-controlled Superiority Trial
Brief Title: Efficacy of Early Argipressin in the Management of Intensive Care Patients With Norepinephrine-refractory Vasoplegic Shock
Acronym: Vaso²R
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGUYEN PHRCN 2023
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Patients With Norepinephrine-refractory Vasoplegic Shock
MeSH Terms: interventions — Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental)
  Interventions: Drug: Argipressin; Other: Collection of clinical data
- Standard group (Active Comparator)
  Interventions: Drug: Chlorure de sodium; Other: Collection of clinical data

INTERVENTIONS:
Drug: Argipressin — Argipressin 0.4 U.ml-1 (i.e. 40IU diluted in 100ml 0.9% NaCl bag)
  Arms: Interventional group
Drug: Chlorure de sodium — NaCl 0.9%
  Arms: Standard group
Other: Collection of clinical data — At inclusion, D0 to D7, ICU discharge, D30 and D90

SUMMARY:
Acute circulatory failure (shock) is defined as insufficient oxygen transport to meet the oxygen requirements of organs and tissues. Vasoplegic shock is the most frequent cause of shock, defined by vasoplegia and a drop in arterial pressure with preserved cardiac output. The main aetiologies of vasoplegic shock are sepsis and post-operative vasoplegia. Symptomatic treatment of vasoplegic shock is based on vasopressors. The first-line vasopressor is norepinephrine. Refractory vasoplegic shock refers as high norepinephrine requirements. In patients with catecholamine-refractory vasoplegia, the use of vasopressin as a second-line treatment is proposed. The use of vasopressin could improve organ and tissue perfusion, improve renal function, accelerate shock reversal and reduce patients' exposure to catecholamines, and thus to their side effects.

Currently, there is a gap between evidence and guidelines/practice regarding vasopressin in patients with refractory vasoplegic shock:

1. There are no large randomized control trial focusing on vasopressin use in patients with refractory vasoplegic shock and data extrapolated from non-refractory shock have contradictory conclusions regarding the benefit of vasopressin in this population.
2. In patients with vasoplegic shock, expert often recommend vasopressin as second line vasopressor and, in the case of septic shock, current international guidelines clearly position vasopressin as second-line therapy in septic shock and advocate its initiation in patients with vasoplegia refractory to norepinephrine.

The strengh of those recommendation is weak due to moderate quality of evidence highlighting the need to conduct a large randomized control trial on this topic.

We hypothesize that the use of vasopressin in patients with refractory vasoplegic shock may improve 30-day survival, decrease renal replacement therapy and reduce duration of vasopressor administration. This is the first multicentred study aiming to confirm the superiority of vasopressin in combination with norepinephrine over norepinephrine alone in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Vasoplegic shock defined as patient requiring vasopressor at the time of inclusion AND with a cardiac index ≥ 2.3/L/min/m² [32] (measured by echocardiography, Swan-Ganz, pulse contour analysis or thermodilution) and with hyperlactatemia > 2 mmol/l.
* Vasoplegia must be primarily caused by one of the following etiologies:

  * Sepsis (documented or clinically suspected infection)
  * Post-operative vasoplegia (following cardiac or non-cardiac surgery)
  * Post hemorrhage
  * Sterile systemic inflammation (e.g., pancreatitis, burns, trauma)
  * Anaphylaxis
  * Liver failure
  * Other causes of vasoplegia
* Refractory shock: dose of vasopressor (express as norepinephrine base equivalent) ≥ 0.25 μg/kg/min in order to maintain perfusion pressure within patient-defined targets (defined by the physician in charge of the patient).
* Early intervention: Criteria for refractory AND vasoplegic shock reached for less than 12 hours.
* Informed consent obtained from the patient or, if unable to give consent, a surrogate. If the surrogate is not available, emergency consent can be considered.
* Covered by French national health insurance

Exclusion Criteria:

* Patients that do not present the criteria for vasoplegic AND refractory shock at the time of inclusion anymore (resolved condition)
* Ongoing vasopressin treatment
* Ongoing inotrope treatment (except norepinephrine)
* Ongoing acute coronary syndrome, mesenteric ischemia
* Uncontrolled active bleeding
* Vasoplegia due to neurogenic shock
* Vasospastic disease (Raynaud's disease, systemic scleroderma…)
* Hyponatremia <120 mmol l-1
* Known hypersensitivity to Argipressin or to any of the excipients of REVERPLEG®.
* Patient already enrolled in an interventional trial
* Decision to limit life-sustaining treatments
* Person under legal protection
* Pregnant, parturient or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
The mortality rate | At Day 30
  in order to determine whether the administration of vasopressin in addition to norepinephrine improves survival
The use of renal replacement therapy within 30 days post-inclusion | At Day 30
  in order to determine whether the administration of vasopressin in addition to norepinephrine improves renal function
The persistence of vasopressor use within 15 days post-inclusion | At Day 15
  to determine whether the administration of vasopressin in addition to norepinephrine reduce the duration of shock

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France